CLINICAL TRIAL: NCT00183209
Title: Interventions for HIV+ Mothers With Problem Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); St. Luke's-Roosevelt Hospital Center (Other); Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAAGWA12113; R01AA012113 (NIH); NIH R01 AA12113
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Substance Use Disorders
Keywords: Substance use disorders; Parent child relationship
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 14 session behavioral intervention (Experimental): 7 sessions addressing problem alcohol and drug use and 7 session addressing parenting challenges (monitoring, negotiation, etc) based on based on Social Action Theory (Ewart, 1991) and Motivational Interviewing
  Interventions: Behavioral: Family First
- Brief Video Intervention (Active Comparator): Single session brief video intervention to build motivation to reduce or eliminate problem drinking/drug use
  Interventions: Behavioral: Family First

INTERVENTIONS:
Behavioral: Family First — Family First = 14 sessions lasting 1.5 hours each based on Social Action Theory and Motivational Interviewing (7 sessions on reducing alcohol and drug use and 7 sessions on reducing parenting challenges). Brief Video Intervention was a single session designed to increase motivation to reduce/eliminate problem drinking or drug use.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a 14-session behavioral intervention for HIV-infected and uninfected mothers with problem drinking. The intervention targets alcohol and drug problems, sexual risk behavior, and parenting. We hypothesize that mothers in the 14-session intervention condition will show improvements in alcohol and drug use, sexual risk behavior, and parenting in comparison to the control condition, which receives a one session brief video intervention.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of a 14-session behavioral intervention for HIV-infected and uninfected mothers with problem drinking. We targeted 118 mothers of adolescent children (aged 11-18). The intervention is based on Social Action Theory (Ewart, 1991) and targets alcohol and drug problems, sexual risk behavior, and parenting. Mothers are followed and interviewed at four intervals over 18 months. Because we anticipate that the intervention will have effects on adolescent behavior, these youth are also enrolled and interviewed at three intervals over 12 months. Adolescents do not attend intervention sessions. We hypothesize that mothers in the 14-session intervention condition will show improvements in alcohol and drug use, sexual risk behavior, and parenting in comparison to the control condition, which receives a one session brief video intervention.

ELIGIBILITY:
Inclusion Criteria for adult participants (mothers):

* Age over 18
* Meets criteria for problem drinking on the AUDIT (score of 6 or greater)
* Has one biological/adopted child aged 11-18 who was in the home at least half the time in the past month

Exclusion Criteria:

* Injection drug use in the past three months

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2001-12; Primary Completion 2006-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Reduction or elimination of alcohol and drug use | 18 months
Reduction or elimination of alcohol/drug use problems | 18 months
Improvement in parenting behaviors (monitoring, communication, etc) | 18 months

SECONDARY OUTCOMES:
Reduction or elimination of sexual risk behavior | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- National Development and Research Institutes, Inc, New York, New York, United States

REFERENCES:
- [Result] Leonard NR, Gwadz MV, Cleland CM, Rotko L, Gostnell K. Physical and mental health functioning of urban HIV-infected and uninfected mothers with problem drinking. Am J Drug Alcohol Abuse. 2007;33(3):419-27. doi: 10.1080/00952990701313652. PMID 17613969
- [Result] de Guzman R, Leonard NR, Gwadz MV, Young R, Ritchie AS, Arredondo G, Riedel M. "I thought there was no hope for me": a behavioral intervention for urban mothers with problem drinking. Qual Health Res. 2006 Nov;16(9):1252-66. doi: 10.1177/1049732306294080. PMID 17038756
- [Result] Gwadz, MV, Leonard, NL, Cleland, C, Riedel, M, Arredondo, G, Wolfe, H, Hardcastle, E, & Morris, J. Behavioral interventions for HIV infected and uninfected mothers with problem drinking. Addiction Research and Theory 16(1): 47-65, 2008.
- [Result] Leonard NR, Gwadz MV, Cleland CM, Vekaria PC, Ferns B. Maternal substance use and HIV status: adolescent risk and resilience. J Adolesc. 2008 Jun;31(3):389-405. doi: 10.1016/j.adolescence.2007.07.001. Epub 2007 Aug 20. PMID 17707902
- [Result] Leonard, N. R., Gwadz, M. V., Arredondo, G. N., Riedel, M., Rotko, L., Hardcastle, E. J., Potere, J. C. (2007). Description of a behavioral intervention to reduce substance use and related risk and increase positive parenting among urban mothers with alcohol and other drug problems. Journal of Child and Family Studies, 16(4):531-544